CLINICAL TRIAL: NCT01436890
Title: A Phase II, 12-week Randomized, Double-blind, Triple Dummy, Parallel Group, Placebo-controlled, Dose Range Finding Study to Evaluate Safety, Tolerability and Efficacy of Revamilast in Patients With Chronic Persistent Asthma
Brief Title: A Clinical Trial to Study the Effects of Revamilast in Patients With Chronic Persistent Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Glenmark Pharmaceuticals Ltd. India (Industry)
Collaborators: Glenmark Pharmaceuticals S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GRC 4039-204; 2011-000270-57 (EudraCT Number)
Record Dates: First submitted 2011-09-14; First posted 2011-09-20 (Estimated); Last update posted 2013-06-21 (Estimated); Status verified 2013-06

CONDITIONS: Asthma
Keywords: Chronic Persistent Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Low dose (Experimental): Low dose revamilast
  Interventions: Drug: Revamilast
- Medium dose (Experimental): Medium dose Revamilast
  Interventions: Drug: Revamilast
- High dose (Experimental): High dose Revamilast
  Interventions: Drug: Revamilast
- Placebo (Placebo Comparator): Matching placebo in triple dummy format
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Revamilast — Tablet. Low dose, Once daily for 12 weeks
  Arms: Low dose
Drug: Revamilast — Medium dose, Once daily for 12 weeks
  Arms: Medium dose
Drug: Revamilast — High dose, Once daily for 12 weeks
  Arms: High dose
Drug: Placebo — Placebo tablet in triple dummy format, Once daily for 12 weeks
  Arms: Placebo

SUMMARY:
Asthma is a common, chronic inflammatory disease of the bronchial airways, with a reported prevalence in most industrialized countries of between 5 to 10 % of the adult population. Asthma is clinically characterized by repeated episodes of wheezing, breathlessness, chest tightness, and coughing; usually in the presence of variable airflow obstruction that is often reversible either spontaneously or with treatment (The Global Initiative for Asthma (GINA), 2009).

Drug treatment of asthma has focused on anti-inflammatory therapy in all but the mildest, intermittent cases. Inhaled corticosteroids have been shown to be anti-inflammatory in asthma, but chronic use of these agents may be associated with a range of side effects, especially at high doses. In asthma, there remains a need for the development of novel anti-inflammatory therapies that are at least equally effective and possess a superior safety profile in comparison to corticosteroids.

This is a randomized, double-blind, triple dummy, placebo controlled, parallel group, dose ranging study. The study will be conducted in adult patients with a diagnosis of chronic persistent asthma with an Forced Expiratory Volume in one second(FEV1) of 50% to 80% of the predicted value. Study will enroll 448 patients globally (278 from India) across different centers.

Patients will be recruited after providing written informed consent. After screening and run in period, patient will be randomized (patient meeting randomization criteria) in 1:1:1:1 ratio to receive either one of the three dose regimens of revamilast or placebo.

The primary objective of the study is to evaluate the effect of revamilast on lung function as assessed by Forced Expiratory Volume in one second (FEV1) after the therapy (12 weeks). Secondary objective includes area under curve for FEV1, Change in asthma symptoms, patient / investigator's global assessments and safety. Patients will be followed for safety and efficacy assessment at week 1, 4, 8 12 and 14 after start of therapy.

ELIGIBILITY:
Inclusion Criteria:

1. The patient provides written informed consent to participate in the study
2. Male or female patient aged 18 to 65 years
3. Documented diagnosis of asthma
4. Forced Expiratory Volume in One Second (FEV1) between 50% and 80% of the predicted value
5. Patient judged by the investigator to be in otherwise good stable health based on medical history, physical examination, and routine laboratory data
6. Female participants must have a negative pregnancy test at screening visit
7. Males must agree to use barrier contraception while on study medication and for 90 days after taking the last dose of study medication

Exclusion Criteria:

1. Pregnant or lactating women
2. Female subjects on hormone replacement therapy or hormonal contraceptives
3. Suffering from relevant lung diseases (other than asthma) causing impairment in lung function
4. Past smoker with a history of ≥10 pack per year or current smoker
5. Recent change in the patient's usual asthma treatment
6. Patients with risk factors for asthma exacerbation during the study, including (any of the following):

   * Current requirement for > 8 puffs per day of reliever medication.
   * Hospitalization for asthma
   * Treatment with systemic corticosteroid therapy within 3 months
7. Evidence of current or recent neoplastic disease
8. Clinically significant cardiovascular, haematological, endocrine, neurological, gastrointestinal, psychiatric, metabolic, immunologic, infectious, hepatic, renal, gynaecological disease or other condition that the investigator considers detrimental to the patient's participation in the study or that may prevent the successful completion of the study
9. Positive serology for an infectious disease (including hepatitis B or C) at screening and known case of human immunodeficiency virus [HIV]
10. Patients who have been hospitalized for any psychiatric illness in the past year, or are diagnosed with major depression
11. Clinically significant ECG Abnormality at baseline
12. Patients with documented or suspected or current history of alcohol and drug abuse
13. Patients who have undergone lung surgery in the previous year
14. Participation in an investigational drug trial during 30 days preceding screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 273 (Actual)
Dates: Start 2011-10; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Change in Forced Expiratory Volume in One Second (FEV1) from baseline to week 12 | Baseline to 12 weeks

SECONDARY OUTCOMES:
Change in morning pre-dose Forced Vital Capacity (FVC) from baseline to week 12 | baseline to 12 weeks
Area under the curve of Forced Expiratory Volume in One Second (FEV1) | 12 weeks
Change in asthma day time symptom score from baseline to week 12 | Baseline to 12 weeks
Frequency and severity of asthma exacerbations during treatment period | 12 weeks
Change in investigator global impression from baseline to week 12 | Baseline to 12 weeks
  An investigator-rated test measured on a 7-point scale, used to rate change in a patient's condition over the course of the study.
Change in patient global impression from baseline to week 12 | Baseline to 12 weeks
  A patient-rated test measured on a 7-point scale, used to rate change in a patient's condition over the course of the study.
Change in morning pre-dose Peak Expiratory Flow (PEF) from baseline to week 12 | Baseline to 12 weeks
Change in morning pre-dose PEF25-75% (Forced expiratory flow 25-75%) from baseline to week 12 | Baseline to 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dr Ballari Brahmachari, Study Director — Glenmark Pharmaceuticals Ltd
Locations (42):
- Czechia (3):
  - HORNMED s.r.o., Brno
  - Sdružená pneumologická a anesteziologická ambulance, Jindřichův Hradec
  - Private pulmonatory ambulance, Neratovice
- India (26):
  - Vasavi Hospital and Research Centre, Hyderabad, Andhra Pradesh
  - Saboo hospital and research centre, Hyderabad, Andhra Pradesh
  - Kunal Institute of Medical Specialities Pvt. Ltd, Hyderabad, Andhra Pradesh
  - Narayana Medical College & Hospital, Nellore, Andhra Pradesh
  - Yashoda Hospital, Secunderabad, Andhra Pradesh
  - T B and Chest Disease Hospital, Mormugao, Goa
  - Rutuja Allergy , Chest and General Clinic, Ponda, Goa
  - Gujarat Pulmonary & Critical Care Clinic, Ahmedabad, Gujarat
  - Chest and Maternity Centre, Bangalore, Karnataka
  - M S Ramaiah Medical College & Teaching Hospital, Bangalore, Karnataka
  - Narayanan Hrudayalaya Hospital, Bangalore, Karnataka
  - Kasturba Medical College Hospital, Mangalore, Karnataka
  - Westfort Hi-tech Hospital Ltd, Thrissur, Kerala
  - Indore Chest Centre, Indore, Madhya Pradesh
  - Prince Aly Khan Hospital, Mumbai, Maharashtra
  - The Bhatia Hospital, Mumbai, Maharashtra
  - KRIMS Hospitals, Nagpur, Maharashtra
  - Getwell Hospital & Research Institute, Nagpur, Maharashtra
  - Chest Research Foundation, Pune, Maharashtra
  - MAMC & Associated Lok Nayak Hospitals, New Delhi, New Delhi
  - Shwaas Center, Navkar Hospital, Jaipur, Rajasthan
  - Asthma Bhawan, Jaipur, Rajasthan
  - Dr Khippal's Clinic, Jaipur, Rajasthan
  - Chennai Thoracic Research Institute, Chennai, Tamil Nadu
  - Christian Medical College, Vellore, Tamil Nadu
  - National Allergy Asthma Bronchitis Institute, Kolkata, West Bengal
- Poland (8):
  - NZOZ 'Promedica', Bialystok
  - Nzoz Clinica Vitae, Gdansk
  - Landa Specjalistyczne Gabinety Lekarskie, Krakow
  - Prywatna Praktyka Lekarska, Krakow
  - Prywatny Gabinet Specjalistyczny, Lodz
  - Cdt Medicus, Lubin
  - Centrum Alergologii Teresa Hofman, Poznan
  - Centrum Medyczne Lucyna Andrzej Dymek, Strzelce Opolskie
- Russia (4):
  - State Healthcare Institution, Elektrostal
  - Central Clinical Hospital of Russian Academy of Science, Moscow
  - State Healthcare Institution of Moscow, Moscow
  - State Educational Healthcare Institution, Saratov
- London Chest Hospital Department of Respiratory Medicine, London, UK, United Kingdom